CLINICAL TRIAL: NCT00962767
Title: A Randomized Study of Two Doses Gemtuzumab Ozogamicin vs. A Two-year Maintenance With Atra Plus Chemotherapy as Post-consolidation Treatment for Intermediate and High-risk Adult Patients With Acute Promyelocytic Leukemia (Apl)
Brief Title: Comparison of Two Treatments in Intermediate and High-risk Acute Promyelocytic Leukemia (APL) Patients to Assess Efficacy in 1st Hematological Complete Remission and Molecular Remission
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0903X-101128
Record Dates: First submitted 2009-08-18; First posted 2009-08-20 (Estimated); Last update posted 2009-08-20 (Estimated); Status verified 2009-08

CONDITIONS: Leukemia, Myelocytic, Acute
Keywords: Oncology comparison study
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Gemtuzumab; Tretinoin; Mercaptopurine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- a (Experimental): 2 doses of gemtuzumab ozogamicn administered at monthly intervals
  Interventions: Drug: gemtuzumab ozogamicin
- b (Active Comparator): 2 years maintenance therapy with intermittent ATRA plus 6-Mercaptopurine (6-MP) and methotrexate (MTX)
  Interventions: Drug: ATRA plus 6-MP and MTX

INTERVENTIONS:
Drug: gemtuzumab ozogamicin — 2 IV infusions 6 mg/m2 administered monthly
  Other Names: Arm A
  Arms: a
Drug: ATRA plus 6-MP and MTX — 6-MP 50 mg/m2/day PO; MTX 15 mg/m2/q week IM; ATRA 45 mg/m2/day PO
  Other Names: Arm B
  Arms: b

SUMMARY:
The study will compare the efficacy of the 2 treatments in intermediate and high-risk APL patients in achieving first hematological complete remission and molecular remission.

ELIGIBILITY:
Inclusion criteria:

1. Patients with untreated newly diagnosed and genetically proven APL (leukemic cells at diagnosis with the t(15;17) and/or the PML/RARα rearrangement by RT-PCR; the presence of additional cytogenetic lesions is not considered an exclusion criterion) with intermediate and high risk disease.
2. Male and female patients age > 18 years and < 61 years.

Exclusion criteria:

1. Low risk patients (WBC < 10 x 109/L and platelets > 40 x 109/L).
2. Absence of PML-RAR α rearrangement in leukemic cells after successful RNA extraction and amplification of control gene.
3. Pretreated APL.

Ages: 18 Years to 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2002-05; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
The study will compare the 2 treatments in intermediate and high-risk APL patients and assess their efficacy in achieving first hematological complete remission and molecular remission. | 5 years

SECONDARY OUTCOMES:
Comparison of short and long-term toxicity of treatment, patient quality of life, and overall survival. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer